CLINICAL TRIAL: NCT02117648
Title: Effects of CYP3A Inhibition by Clarithromycin on the Pharmacokinetics of LY2835219 and Its Metabolites in Cancer Patients
Brief Title: A Study of LY2835219 in Participants With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15173; I3Y-MC-JPBE (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Neoplasm; Neoplasm Metastasis
Keywords: advanced cancer; metastatic cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — abemaciclib; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abemaciclib Alone Period 1 (Experimental): 50 mg single oral dose of Abemaciclib was administered in Period 1 Day 1.
  Interventions: Drug: Abemaciclib
- Abemaciclib + Clarithromycin Period 2 (Experimental): Clarithromycin 500 milligram (mg) orally twice daily for 12 days. Single oral dose of Abemaciclib 50 mg on Period 2 Day 5. Clarithromycin dosing continued for 7 days following the single dose of Abemaciclib.
  Interventions: Drug: Abemaciclib; Drug: Clarithromycin
- Abemaciclib Safety Extension (Experimental): After completing Period 2, eligible participants continued to receive 200 mg Abemaciclib every 12 hours (Q12H) on a 28-day cycle in a safety-extension phase until discontinuation criteria were met.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Clarithromycin — Administered orally
  Arms: Abemaciclib + Clarithromycin Period 2

SUMMARY:
The purpose of this study is to assess how the body handles Abemaciclib when it is given with another drug called clarithromycin. The study doctor will measure the amount of Abemaciclib that is absorbed into the blood stream and the time that it takes to remove Abemaciclib from the body. The safety and tolerability of these drugs will be studied.

Each participant will complete 2 study periods in fixed order. After screening, Period 1 will last approximately 8 days and Period 2 will last approximately 15 days. Participants who complete Period 2 may continue to receive Abemaciclib in 28-day cycles until discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of cancer (solid tumors) that is advanced and/or metastatic
* Have a performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) scale

Exclusion Criteria:

* No symptomatic central nervous system (CNS) malignancy or metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Accelerated Comm. Oncology Research Network (ACORN), Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee

REFERENCES:
- [Derived] Gelbert LM, Cai S, Lin X, Sanchez-Martinez C, Del Prado M, Lallena MJ, Torres R, Ajamie RT, Wishart GN, Flack RS, Neubauer BL, Young J, Chan EM, Iversen P, Cronier D, Kreklau E, de Dios A. Preclinical characterization of the CDK4/6 inhibitor LY2835219: in-vivo cell cycle-dependent/independent anti-tumor activities alone/in combination with gemcitabine. Invest New Drugs. 2014 Oct;32(5):825-37. doi: 10.1007/s10637-014-0120-7. Epub 2014 Jun 13. PMID 24919854

RESULTS

PARTICIPANT FLOW:
Groups:
- Abemaciclib Alone Then Abemaciclib + Clarithromycin: 50 mg single oral dose of Abemaciclib was administered on Period 1 Day 1 and on Period 2 Day 5. Clarithromycin 500 milligram (mg) orally twice daily for 12 days. Clarithromycin dosing continued for 7 days following the single dose of Abemaciclib. After completing Period 2, eligible participants continued to receive 200 mg Abemaciclib every 12 hours (Q12H) on a 28-day cycle in a safety-extension phase until discontinuation criteria were met.
Period: Abemaciclib Alone Period 1
Arm/Group | Abemaciclib Alone Then Abemaciclib + Clarithromycin
Started | 26
Received at Least 1 Dose of Study Drug | 26
Completed | 24
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Period: Abemaciclib + Clarithromycin Period 2
Arm/Group | Abemaciclib Alone Then Abemaciclib + Clarithromycin
Started | 24
Received at Least 1 Dose of Study Drug | 21
Completed | 20
Not Completed | 4
Not completed — Progressive Disease | 1
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Abemaciclib Safety-Extension Phase
Arm/Group | Abemaciclib Alone Then Abemaciclib + Clarithromycin
Started | 20
Completed | 0
Not Completed | 20
Not completed — Progressive Disease | 12
Not completed — Physician Decision | 1
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Abemaciclib Then Abemaciclib + Clarithromycin: 50 mg single oral dose of Abemaciclib was administered on Period 1 Day 1 and on Period 2 Day 5. Clarithromycin 500 mg orally twice daily for 12 days. Clarithromycin dosing continued for 7 days following the single dose of Abemaciclib. After completing Period 2, eligible participants continued to receive 200 mg Abemaciclib Q12H on a 28-day cycle in a safety-extension phase until discontinuation criteria were met.
Arm/Group | Abemaciclib Then Abemaciclib + Clarithromycin
Number analyzed (Participants) | 26
Age, Customized [Mean (Standard Deviation); unit: years] | 60.0 (9.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 19
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/square meter (kg/m2)] | 27.62 (6.04)
Eastern Cooperative Oncology Group (ECOG) Scale [Number; unit: participants] — ECOG 0 = Fully active, able to carry on all predisease performance without restriction
  ECOG 1 = Restricted in physically strenuous activity but ambulatory and able to carry out performance of a light or sedentary nature, for example, light housework, office work
  participants
    ECOG= 0 | 18
    ECOG= 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Zero to Infinity (AUC[0-∞]) of Abemaciclib
Time Frame: Period 1: Predose; 1, 2, 4, 6, 8, 10, 24, 48, 72, 96, 120, 144, 168hr, Period 2: 1, 2, 4, 6, 8, 10, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240hr Post dose
Population: All participants who received at least 1 dose of study drug and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter(mL) ng*h/mL
Groups:
- Abemaciclib Period 1: 50 mg single oral dose of Abemaciclib was administered in Period 1 Day 1.
- Abemaciclib + Clarithromycin Period 2: Starting on Period 2 Day 1, Clarithromycin 500 mg orally twice daily for 12 days. Single oral dose of Abemaciclib on Period 2 Day 5. Clarithromycin dosing continued for 7 days following the single dose of Abemaciclib.
Arm/Group | Abemaciclib Period 1 | Abemaciclib + Clarithromycin Period 2
Number analyzed (Participants) | 26 | 19
nanogram*hour/milliliter(mL) ng*h/mL | 2230 (93) | 6850 (66)

2. Primary Outcome: PK: Maximum Concentration (Cmax) of Abemaciclib
Time Frame: Period 1: Predose; 1, 2, 4, 6, 8, 10, 24, 48, 72, 96,120,144,168hr, Period 2: 1, 2, 4, 6, 8, 10, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240hr Post dose
Population: All participants who received at least 1 dose of study drug and had evaluable cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Abemaciclib Period 1 | Abemaciclib + Clarithromycin Period 2
Number analyzed (Participants) | 26 | 19
nanogram/milliliter (ng/mL) | 70.0 (73) | 84.3 (55)

ADVERSE EVENTS:
Groups:
- Abemaciclib: 50 mg single oral dose of Abemaciclib was administered in Period 1 Day 1.
- Clarithromycin: Clarithromycin 500 mg orally twice daily for 12 days
- Abemaciclib + Clarithromycin: Clarithromycin 500 mg orally twice daily for 12 days. Single oral dose of Abemaciclib on Period 2 Day 5 . Clarithromycin dosing continued for 7 days following the single dose of Abemaciclib.
- Safety Extension Abemaciclib: After completing Period 2, eligible participants continued to receive 200 mg Abemaciclib Q12H on a 28-day cycle in a safety-extension phase until discontinuation criteria were met.
Arm/Group | Abemaciclib | Clarithromycin | Abemaciclib + Clarithromycin | Safety Extension Abemaciclib
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/24 | 1/21 | 15/20
Other Adverse Events (participants affected / at risk) | 13/26 | 7/24 | 10/21 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=26) | Clarithromycin (N=24) | Abemaciclib + Clarithromycin (N=21) | Safety Extension Abemaciclib (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Abemaciclib (N=26) | Clarithromycin (N=24) | Abemaciclib + Clarithromycin (N=21) | Safety Extension Abemaciclib (N=20)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2) | 12 (15)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 12 (17)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 9 (12)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 7 (11)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 14 (19)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Vaginal infection (Infections and infestations) | 0/19 (0) | 0/19 (0) | 0/17 (0) | 1/16 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 8 (10)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 9 (17)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/19 (0) | 0/19 (0) | 0/17 (0) | 1/16 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days